CLINICAL TRIAL: NCT06569810
Title: Real-world Registry Study of Red Light Treatment on Myopia Control: a Focus on Non-responders to Conventional Treatments
Status: Not yet recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Other Study IDs: HSEARS20240113001
Record Dates: First submitted 2024-08-05; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-04

CONDITIONS: Myopia; Repeated Low-level Red Light
MeSH Terms: conditions — Myopia | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-responders to Conventional Treatments: This observational, real-world, web-based registry study will collect treatment data from multiple clinics of children aged 8-16 years old who have insufficient control of progression under myopia treatments for at least six months, and are receiving or intend to receive RLRL therapy. Insufficient control is defined as meeting either of the following criteria: AL elongation of less than 0.3mm per year or SER progression of 0.5 diopter (D) or greater per year. These subjects will then be defined as non-responders to conventional treatments for myopia, and offered RLRL therapy.
  Interventions: Device: Repeated Low-Level Red Light (RLRL) therapy

INTERVENTIONS:
Device: Repeated Low-Level Red Light (RLRL) therapy — In our study, we do not implement any interventions; rather, we collect follow-up information from patients who, due to insufficient response to traditional myopia control therapies, have transitioned to Repeated Low-Level Red Light (RLRL) therapy. The data gathered will reflect treatment patterns as per the approved indications for RLRL therapy, where subjects may have undergone treatment sessions twice daily, each lasting for 3 minutes with a minimum interval of 4 hours between sessions. Our analysis will focus on the real-world outcomes, specifically evaluating the proportion of participants who have achieved effective myopia control (defined as AL elongation of less than 0.1mm per year or SER progression of less than 0.25 diopter per year) after 12 months of documented RLRL therapy use among the collected data from eligible subjects.

SUMMARY:
This real-world observational registry study aims to assess the effectiveness of Repeated Low-Level Red Light (RLRL) therapy in controlling myopia progression among children aged 8 to 16 who have not responded to conventional treatments like Orthokeratology and atropine eyedrops. The primary focus is to determine if RLRL therapy can limit axial length (AL) elongation to less than 0.1mm per year and spherical equivalent refraction (SER) progression to less than 0.25 diopter per year, while also evaluating safety and visual outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 8 to 16 years at the time of data collection, aligning with the approved usage guidelines of the RLRL device.
2. Diagnosed with myopia and have been under conventional myopia treatments (include Orthokeratology, defocus incorporated multiple segments spectacles or equivalent, and 0.01% atropine or 0.05% atropine eyedrops) for at least six months. Eligible patient data must demonstrate insufficient control of myopia progression, defined as an axial elongation of 0.3 mm or more, or SER progression of 0.5 diopter or greater per year.
3. Best corrected visual acuity (BCVA): 20/20 or greater.
4. Data from patients who have utilized or are utilizing red light therapy as part of their myopia management strategy.

Exclusion Criteria:

1. Ophthalmic diseases other than refractive errors, including but not limited to strabismus and binocular vision abnormalities in either eye.
2. Presence of systemic diseases (e.g., endocrine, cardiac diseases) and developmental abnormalities.
3. Concurrent use of atropine eye drops and RLRL therapy.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The design of our study as a data registry project fundamentally shapes our approach to sample size estimation. Unlike traditional clinical trials, our study does not involve experimental interventions but instead collects real-world clinical data from patients on RLRL therapy. Consequently, our sample size will reflect the number of patients treated with RLRL in participating clinics during the study period. We anticipate significant uptake of this therapy, aiming to recruit up to 2,500 participants within one year, given its approval and present adoption in clinical practice. This estimated amount of participation is likely to provide a robust sample size, enhancing the statistical power and generalizability of our findings.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of fully controlled | 12 months for each participate
  The proportion of the people with AL elongation of less than 0.1mm per year or SER progression of less than 0.25 diopter per year after RLRL therapy for 12 months.

SECONDARY OUTCOMES:
BCVA changes | 12 months for each participate
  Best corrected visual acuity (BCVA) changes at 12 months.
Optical coherence tomography (OCT) scan changes (eg. choroidal thickness changes on OCT scans.) | 12 months for each participate
  Optical coherence tomography (OCT) scan changes at 12 months.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT06569810/ICF_000.pdf